

# Modified Vascularized Interpositional Periosteal Connective Tissue Graft Versus Xenogeneic Collagen Matrix For soft tissue Augmentation Around Implant in Esthetic Zone (A Comparative Study)

Proposal

Presented By

Heba Ahmed Abd El-Maged Elsweefy

25/12/2024

### **Statistical Analysis:**

Statistical analysis was performed with IBM® SPSS® (ver. 26. SPSS Inc., IBM Corporation, Armonk, NY, USA). Data explored for normality using Shapiro-Wilk test. Quantitative data were presented by mean and standard deviation. Independent t test was used to compare means between two groups. Paired t test was used to compare between two means before and after treatment within each group. A repeated measure ANOVA is used to compare means in each group across multiple times to see changes to an intervention. A statistically significant level was considered when p value < 0.05.

#### 3. Results:

Twenty patients were recruited in the study, including 12 females and 8 males aged between 20 to 40 years; there were no failed implants or withdrawal of any patients during the follow-up period. Every one of the participants had their planned treatment, and all the implants placed osseointegrated successfully. Data are expressed as mean  $\pm$  standard deviation.

#### 3.1 Clinical Parameters:

- **3.1.1 keratinized tissue thickness:** KTT increased from baseline to 3, 6 months in both of groups but more improvement seen in mVIP-CT group than in XCM group at 3 and 6 month. No significant differences between the study groups at baseline, but at 3 and 6 month the differences were statistically significant
- **3.1.2 keratinized tissue width:** KTW increased from baseline to 3,6 months in both groups but was slightly higher in mVIP-CT group than in XCM group at 6 months with nonsignificant differences between them at baseline and follow up
- **3.1.3 pink esthetic score:** The aesthetic outcome was measured by Pink Esthetic Score (PES), the comparison between both groups revealed a non-significantly higher results in mVIP-CT group than in XCM group

## 3.2. Radiographic Parameters:

**3.2.1 buccal cortex thickness**: increased from baseline to 6 month in both of mVIP-CT group and XCM group with no significant differences between the study groups at baseline and follow up period.

Table (1): Keratinized tissue thickness (KTT) level at different points of time in mVIP-

CTG group

| KTT | n | VIP-CTG group P value Baseline | | P value<br>Baselin | P value | |
|---|---|---|---|---|---|---|
| | Baseline | 3<br>months | 6 months | vs<br>3 months | e vs<br>6<br>months | months<br>vs<br>6 |
| | | | | | | months |
| Mean±SD | 1.5±0.53 | 1.9±0.41 | 2.8±0.56 | 0.9 | 0.001* | 0.01* |

Table (2): Keratinized tissue thickness (KTT) level at different points of time in XCM

group

| KTT | 8 1 | | | | P value<br>3 months | |
|---|---|---|---|---|---|---|
| | Baseline | 3 months | 6 months | vs<br>3<br>months | vs<br>6<br>months | vs<br>6 months |
| Mean±SD | $1.4 \pm 0.67$ | 1.5±0.40 | 2.0±0.55 | 0.1 | 0.2 | 0.5 |



Table (3): Keratinized tissue thickness (KTT) level between groups

| KTT | Groups | P value | |
|-------------|-----------------|--------------|-------|
| | mVIP-CTG (n=10) | XCM (n=10) | |
| | Mean±SD | Mean±SD | |
| At baseline | 1.5±0.53 | 1.4±0.67 | 0.7 |
| 3 months | 1.9±0.41 | 1.5±0.40 | 0.04 |
| 6 months | 2.8±0.56 | $2.0\pm0.55$ | 0.004 |



Table (4): Keratinized tissue width (KTW) level at different points of time in mVIP-

CTG group

| KTW | mVIP-CTG group | | | P value<br>Baseline | P value 3 | |
|---|---|---|---|---|---|---|
| | Baselin<br>e | 3 months | 6<br>months | vs<br>3<br>months | vs<br>6<br>months | months<br>vs<br>6 |
| | | | | | | months |
| Mean±SD | 1.4±0.52 | 1.5±0.53 | 2.0±0.84 | 0.9 | 0.07 | 0.1 |

Table (5): Keratinized tissue width (KTW) level at different points of time in XCM group

| KTW | | XCM group | | P value<br>Baseline | P value<br>Baseline | P value<br>3 months |
|---|---|---|---|---|---|---|
| | Baseline | 3 months | 6 months | vs<br>3 months | vs<br>6 | vs<br>6 months |
| | | | | | months | |
| Mean±SD | 1.6±0.52 | 1.7±0.52 | 1.9±0.68 | 0.6 | 0.2 | 0.4 |



Table (6): Keratinized tissue width (KTW) level between groups

| KTW | Groups | P value | |
|-------------|-----------------|--------------|-----|
| | mVIP-CTG (n=10) | XCM (n=10) | |
| | Mean±SD | Mean±SD | |
| At baseline | 1.4±0.52 | 1.6±0.52 | 0.3 |
| 3 months | 1.5±0.53 | $1.7\pm0.52$ | 0.4 |
| 6 months | 2.0±0.84 | $1.9\pm0.68$ | 0.7 |



Table (7): Buccal cortex thickness level at baseline and after 6 months in mVIP-CTG

group

| Buccal cortex<br>thickness | mVIP-CTG group | | Mean<br>differenc | P value |
|---|---|---|---|---|
| <b>CARCALLO</b> SS | Baseline | 6 months | e | |
| Mean±SD | 0.744±0.33 | 1.207±0.16 | -0.463 | 0.01 |



Table (8): Buccal cortex thickness level at baseline and after 6 months in XCM group

| Buccal cortex<br>thickness | XCM group | | 8 1 | | Mean<br>differenc | P value |
|---|---|---|---|---|---|---|
| | Baseline | 6 months | e | | | |
| Mean±SD | $0.92 \pm 0.32$ | 0.97±0.31 | -0.054 | 0.6 | | |



Table (9): Buccal cortex thickness level between groups

| <b>Buccal cortex thickness</b> | Groups | P value | |
|---|---|---|---|
| | mVIP-CTG (n= 10) XCM (n=10)<br>Mean±SD Mean±SD | | |
| At baseline | 0.744±0.33 | 0.92±0.32 | 0.2 |
| 6 months | 1.207±0.16 | $0.97 \pm 0.31$ | 0.06 |



Table (10): Pink esthetic score (PES) between groups

| | Group | P value | |
|---|---|---|---|
| | mVIP-CTG (n= 10)<br>Mean±SD | XCM (n=10)<br>Mean±SD | |
| Pink esthetic score (PES) | 6.8±0.57 | 6.3±0.53 | 0.06 |

